CLINICAL TRIAL: NCT04962893
Title: Phase II Study to Assess the Safety, Efficacy, and Immunogenicity of Authentic SARS-CoV-2 or Alpha Variant Spike Containing VLP Vaccines and Their Combination for the Prevention of COVID-19 in Healthy Adult Volunteers (SAVE STUDY)
Brief Title: Study of a Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Virus-like Particle (VLP) Vaccine
Acronym: COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ihsan GURSEL, PhD, Prof. (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Nobel Pharmaceuticals (Industry); MonitorCRO (Industry)
Responsible Party: Sponsor-Investigator, Ihsan GURSEL, PhD, Prof., Co- Principal Investigator, The Scientific and Technological Research Council of Turkey
Organization: The Scientific and Technological Research Council of Turkey (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VLP-58-1023-Al-K3-PII
Record Dates: First submitted 2021-07-12; First posted 2021-07-15 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Covid19
Keywords: Virus-like Particles harboring S, M, N, E antigens; SARS-CoV-2; K3-CpG ODN; Alum
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VLP-Wuhan group (Group V1) (Experimental): 110 participants will receive 40 mcg of Alum adsorbed VLP vaccine for Wuhan adjuvanted with K3-CpGODN (1 ml), in two doses 21 days apart.
  Interventions: Biological: SARS-CoV-2 VLP Vaccine-Wuhan
- VLP-Alpha (British) variant group (Group V2) (Experimental): 110 participants will receive 40 mcg of Alum adsorbed VLP vaccine for Alpha variant adjuvanted with K3-CpGODN (1 ml), in two doses 21 days apart.
  Interventions: Biological: SARS-CoV-2 VLP Vaccine-Alpha (British) variant
- VLP-Wuhan+Alpha group (Group V3) (Experimental): 110 participants will receive 40 mcg of Alum adsorbed VLP vaccine for Wuhan and Alpha variant adjuvanted with K3-CpGODN (1 ml), in two doses 21 days apart.
  Initial vaccination with Wuhan followed by a booster of Alpha variant.
  Interventions: Biological: SARS-CoV-2 VLP Vaccine-Wuhan+Alpha variant

INTERVENTIONS:
Biological: SARS-CoV-2 VLP Vaccine-Wuhan — Alum adsorbed, CpG ODN adjuvanted VLP vaccine expressing HexaPro-S, M, N, E proteins of the virus
  Other Names: Authentic VLP Vaccine
  Arms: VLP-Wuhan group (Group V1)
Biological: SARS-CoV-2 VLP Vaccine-Alpha (British) variant — Alum adsorbed, CpG ODN adjuvanted VLP vaccine expressing HexaPro-S, M, N, E proteins of the virus
  Other Names: Alpha Variant VLP Vaccine
  Arms: VLP-Alpha (British) variant group (Group V2)
Biological: SARS-CoV-2 VLP Vaccine-Wuhan+Alpha variant — Alum adsorbed, CpG ODN adjuvanted VLP vaccine expressing HexaPro-S, M, N, E proteins of the Wuhan or Alpha variants
  Other Names: Combination of Authentic and Alpha VLP Vaccine
  Arms: VLP-Wuhan+Alpha group (Group V3)

SUMMARY:
This is a randomized, parallel dose assigned, double blind, multi center, Phase II study assessing the efficacy, safety, and immunogenicity of VLP vaccine (Authentic and Alpha variants) in adults between 18 and 59 years who are healthy or have medically stable chronic diseases and who have no known history of SARS-CoV-2 infection

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the humoral and cellular immune response of VLP vaccine candidates (harboring M, N, E, and HexaPro S antigens of the virus), as an efficacy criteria.

Approximately 330 subjects will be randomized in a 1:1:1 ratio to receive two doses of 40 mcg VLP vaccine for Wuhan (n=110) or 40 mcg VLP vaccine for Alpha (British) variant (n=110) or 40 mcg VLP vaccine for Wuhan+Alpha variant (n=110) 21 days apart.

The study will be completed in 14 months.

All injections will be done subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, each participant must satisfy all the following criteria:

1. Female and/or male participant who is informed and about his/her participation and who agrees to give his/her written informed consent.
2. Aged between 18 and 59 years.
3. Negative Immunoglobulin G (IgG)/Immunoglobulin M (IgM) antibody for COVID-19.
4. Negative COVID-19 quantitative polymerase chain reaction (qPCR) test result.
5. Able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
6. Negative blood test for hepatitis B (HBV), hepatitis C (HCV) and human immunodeficiency virus (HIV) at screening period.
7. Body temperature < 37.2°C.
8. Body Mass Index (BMI) ranged between 18-35 kg/m2.
9. Clinical laboratory test results within the reference range of the laboratory or clinically non-significant (complete blood count (CBC), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, urea, creatinine, and fasting glucose) or any laboratory parameters defined in the study protocol.
10. Good general health as determined by physical examination, laboratory screening, and review of medical history within 14 days prior to participation.
11. Female participants of childbearing potential may be enrolled in the study if the subject fulfils all the following criteria:

    * Have a negative pregnancy test on the day of screening and prior to each study vaccine administration.
    * Use an effective contraceptive method for at least 30 days prior to first dose of study vaccine and agree to continue using one highly effective form of birth control through 6 months after the administration of the last dose of study vaccine.
12. Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as postmenopausal (defined as amenorrhea for ≥12 consecutive months prior to Screening without an alternative medical cause) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
13. Male participants who agree to use an effective contraceptive method during the study period and until 6 months after the last dose of study vaccine.

Exclusion Criteria:

Participants with any of the following criteria will be excluded:

1. History of laboratory-confirmed SARS-COV-2 infection.
2. History of seizures, encephalopathy, or psychosis.
3. Known or suspected allergy or history of anaphylaxis or other serious adverse reactions to any vaccine or study vaccine and/or any other excipients of the vaccine.
4. Pregnant, breastfeeding or planning to become pregnant within 6 months after the study vaccine administration.
5. Suspected active infection or other acute illness, including fever > 37.2°C.
6. Any presence of clinical relevance of cardiovascular disease (including but not limited to arrythmia, myocardial infarction, uncontrolled hypertension, coronary artery disease, or congestive heart failure).
7. Any presence of clinical relevance of serious chronic disease [asthma, diabetes, thyroid diseases etc.).
8. Any presence of clinical relevance of congenital or acquired angioedema.
9. Diagnosis of immunodeficiency.
10. Diagnosis of bleeding diathesis.
11. Use of immunosuppressive medications, anti-allergic therapy, cytotoxic therapy, inhaler corticosteroids (excluding allergic rhinitis or topical steroid ointments).
12. Those who received blood/plasma products or immunoglobulins and/or blood transfusion within the last 6 months.
13. Those who participated in another vaccine study or received an investigational/experimental drug within 1 month prior to study entry.
14. History of any live vaccine within 1 month prior to study participation.
15. History of any inactivated vaccine within 1 month prior to study participation.
16. Use of active tuberculosis treatment.
17. According to the investigator's judgement, those who have any condition (medical, psychological, social, etc.) that may impair the subject's compliance with the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 349 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
Comparison of efficacy | On Day 14 after booster dose administration
  Comparison of antibody responses of participants to a cohort of standard convalescent serum samples obtained from World Health Organization (WHO).
Comparison of efficacy | On Day 28 after booster dose administration
  Comparison of antibody responses of participants to a cohort of standard convalescent serum samples obtained from World Health Organization (WHO).
Specific antibody (IgG) response | On Day 14 after booster dose administration
  SARS-CoV-2 Spike/S1 or RBD antibody titers
Specific antibody (IgG) response | On Day 28 after booster dose administration
  SARS-CoV-2 Spike/S1 or RBD antibody titers
Neutralizing antibody response | On Day 14 after booster dose administration
  Neutralizing antibody titer against anti-Spike protein by virus neutralization method developed against SARS-CoV-2
Neutralizing antibody response | On Day 28 after booster dose administration
  Neutralizing antibody titer against anti-Spike protein by virus neutralization method developed against SARS-CoV-2
Cellular immune response | Before first dose administration, on Day 14 after booster dose administration
  ELISPOT: Interferon-γ (IFN-γ) positive level of T-cells

SECONDARY OUTCOMES:
Adverse events (AEs) | Until Month 12 after booster dose administration
  Local and systemic AEs in all vaccine groups
Serious adverse events (SAEs) | Until Month 12 after booster dose administration
  SAEs in all vaccine groups
Specific antibody (IgG) response | Before first and booster dose administration, at Month 3, Month 6, Month 9 and Month 12 after booster dose
  SARS-CoV-2 Spike/S1 or RBD antibody titers

CONTACTS AND LOCATIONS:
Overall Officials: Fevzi ALTUNTAS, Principal Investigator — HEAD OF ONCOLOGY HOSPITAL
Locations (3):
- Turkey (Türkiye) (3):
  - Dr. Abdurahman Yurtaslan Ankara Oncology Training and Research Hospital Phase I Clinical Study Center, Ankara
  - Health Sciences University İstanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul
  - Kocaeli University Research and Application Hospital Infectious Disease and Clinical Microbiology Department, Kocaeli

REFERENCES:
- [Derived] Yilmaz IC, Ipekoglu EM, Golcuklu BS, Bildik T, Aksoy AGB, Evcili I, Turay N, Surucu N, Bulbul A, Guvencli N, Yildirim M, Canavar Yildirim T, Atalay YA, Abras I, Ceylan Y, Ozsurekci Y, Tigen ET, Korten V, Gursel M, Gursel I. A phase I/II study of CpG/alum-adjuvanted mammalian-derived quadruple antigen carrying virus-like particle COVID-19 vaccine. Vaccine. 2025 Mar 7;49:126787. doi: 10.1016/j.vaccine.2025.126787. Epub 2025 Jan 31. PMID 39892108